CLINICAL TRIAL: NCT00299585
Title: Phase 2 Clinical Study on the Efficacy of Injectable Brushite Bone Cement in Bone Augmentation and Dental Implant Stabilization
Brief Title: A Clinical Study of the Use of Brushite as Primary Stabilizer in Immediate Dental Implantation
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: manufacturer could not finance the study
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arik Tzukert, DMD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 191059 HMO-CTIL
Record Dates: First submitted 2006-03-05; First posted 2006-03-07 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2007-12

CONDITIONS: Alveolar Ridge Augmentation; Dental Implants
Keywords: dental implant; dental implantation; osseointegration; bone cement; osteoconductivity; brushite; calcium phosphate; bone augmentation; primary stability; immediate implantation; Mandibular Ridge Augmentation; Maxillary Ridge Augmentation; synthetic implants for rebuilding the alveolar ridge
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: using "PD" VitalOs Cement with dental implants — supporting dental implants with Vitalos bone cement

SUMMARY:
Objective: The evaluation of "PD" VitalOs Cement, an injectable brushite, as a stabilizer of dental implants and a potential source for bone augmentation.

Methods: Forty (40) patients needing dental implants will be treated where needed with "PD" VitalOs Cement gapping half of their sites whereas the other half will be gapped with Bio-oss demineralized bone and BioGuide membrane.

DETAILED DESCRIPTION:
Bone fractures or bone loss in specific sites are cases where a bone graft is sometimes needed to provide bone augmentation. For bone fractures, these are typically metaphyseal or maxillofacial fractures with risk of malunion or non-union. Bone loss can happen under various circumstances: it can be a consequence of a systemic disease like osteoporosis or of a surgical intervention like the extraction of a tooth or the removal of a bone cyst or tumor.

When a bone graft is required the gold standard still widely used is autogenous cancellous bone. However, the graft harvesting procedure is invasive and increases patient morbidity (lengthened surgical procedure, increased risk of infection). Moreover, the availability of autologous grafts is limited, especially in elderly patients. This has been the rationale for studying alternative sources for bone grafts.

The first alternative is allografts: they are usually obtained from cadavers. The advantages include elimination of a patient donor site, hence reduced surgical time and decreased blood loss and risk of infection. The principal shortcomings are the availability, the possible rejection of the graft and the risk of disease transmission.

Grafts of animal origin (xenografts) are also an option, even though not totally risk-free when it comes to disease transmission.

A third alternative to autologous bone is to use synthetic materials. Extensive research has been performed to develop such materials since the 80's. The majority of them are based on calcium phosphate compounds, made up of the same ions as those of the natural mineral phase of bone. These products are readily available, eliminate the risk of disease transmission or immunogenic response (allografts) and bypass the need for an additional surgical procedure (autografts). These materials are presented under either of the three forms: granules, pre-formed blocks or cements.

Granules and pre-formed blocks are generally made up of β-TCP, Hydroxyapatite (HA), or a mix of both. Depending mainly on their chemical composition, their manufacturing process and their porosity, they degrade more or less rapidly.

Calcium phosphate cements consist generally of a liquid and a powder which harden upon mixing. The final product phase can be hydroxyapatite, or another calcium phosphate phase like dahllite or brushite. The advantage of cements over pre-formed blocks is that they can be injected, shaped and hardened in situ, ensuring optimum bone-implant contact and minimally invasive surgery. Once hardened, they exhibit cohesive properties that granules cannot provide. Most of the calcium phosphate cements available on the market are hydroxyapatite cements. However, for some applications like periodontitis or peri-implant gap filling, their resorption rate is too slow, hampering their clinical applicability for these indications. The advantage of the brushite phase in the hardened cement is that it degrades faster than hydroxyapatite, allowing a more rapid bone regeneration. The purpose of this study is to evaluate the efficacy of "PD" VitalOs Cement as a primary stabilizer and bone augmenting source in dental implantology.

ELIGIBILITY:
Inclusion Criteria:

* Partially or fully edentulous patients who need dental implants to support a prosthesis

Exclusion Criteria:

* Patients with uncontrolled diabetes
* Chemotherapy
* Immune suppressed
* Radiotherapy to head and neck in the last five years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
X-ray evaluation of osseointegration | 3-6 12 months
clinical assesment | 3-6 and12

SECONDARY OUTCOMES:
long-term follow-up for osseointegration: clinical and X-ray | 12-18-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Perez Davidi, DMD, Study Chair — Hadassah Medical Organization; Nardi Caspi, DMD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Background] Pittet C, Lemaitre J. Mechanical characterization of brushite cements: a Mohr circles' approach. J Biomed Mater Res. 2000;53(6):769-80. doi: 10.1002/1097-4636(2000)53:63.0.co;2-p. PMID 11074436
- [Result] Charriere E, Terrazzoni S, Pittet C, Mordasini PH, Dutoit M, Lemaitre J, Zysset PH. Mechanical characterization of brushite and hydroxyapatite cements. Biomaterials. 2001 Nov;22(21):2937-45. doi: 10.1016/s0142-9612(01)00041-2. PMID 11561900
- See also: Michael Perez Davidi — http://www.mypd.co.il